CLINICAL TRIAL: NCT00912444
Title: A Multi-Center, Randomized Study of Docetaxel, Anthracycline and Cyclophosphamide (TAC) Versus Docetaxel and Cyclophosphamide (TC) in Neoadjuvant Treatment of Triple-Negative or Her2 Positive Breast Cancer
Brief Title: Neoadjuvant Treatment of Docetaxel, Anthracycline and Cyclophosphamide (TAC) Versus Docetaxel and Cyclophosphamide (TC) in Triple-Negative or Her2 Positive Breast Cancer
Acronym: NATT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: TAC treatment was associated with better survial outcome compared with TC treatment, we terminated recruiting and waiting for longer follow up period.
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NATT
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
Keywords: Breast Neoplasms; Neoadjuvant; Chemotherapy; Docetaxel; Cyclophosphamide; Anthracycline
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Anthracyclines; Doxorubicin; Epirubicin; Cyclophosphamide; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAC Arm (Experimental): six cycles of neoadjuvant Docetaxel, Anthracycline and Cyclophosphamide
  Interventions: Drug: Docetaxel, Anthracycline (Doxorubicin or Epirubicin), Cyclophosphamide
- TC Arm (Experimental): six cycles of neoadjuvant Docetaxel and Cyclophosphamide
  Interventions: Drug: Docetaxel, cyclophosphamide

INTERVENTIONS:
Drug: Docetaxel, Anthracycline (Doxorubicin or Epirubicin), Cyclophosphamide — Docetaxel 75mg/m2, doxorubicin 50mg/m2 or epirubicin 60mg/m2, cyclophosphamide 500mg/m2 every 3 weeks for six cycles
  Arms: TAC Arm
Drug: Docetaxel, cyclophosphamide — Docetaxel 75mg/m2, cyclophosphamide 600mg/m2 every 3 weeks for six cycles
  Arms: TC Arm

SUMMARY:
The purpose of this study is to compare the pathological complete response (pCR) rate in triple-negative or Her2 positive breast cancer patients treated with neoadjuvant docetaxel, anthracycline and cyclophosphamide (TAC) or docetaxel and cyclophosphamide (TC) regimen.

DETAILED DESCRIPTION:
Breast cancer is the leading cause of cancer in women in China. Neoadjuvant chemotherapy for treatment of locally advanced breast cancer has become a standard therapy. Results from neoadjuvant trials have shown that pathological complete response (pCR) is an independent predictor of outcome. Docetaxel was introduced into clinical practice in the early 1990s and has demonstrated good activity in the adjuvant and metastatic settings. Both TC and TAC are effective regimens in the adjuvant setting. The most optimal regimen in the neoadjuvant treatment is however unknown. This is especially true in triple-negative or HER2 positive breast cancer. This study will evaluate the pCR rate of TAC and TC as neoadjuvant treatment for triple-negative or HER2 positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years and < 70 years
* Karnofsky performance status (KPS) ≥ 70
* At least one measurable disease according to the RECIST. histologically confirmed invasive breast cancer (excluding inflammatory breast cancer), T2N1 or locally advanced breast cancer (T3-4N0-3 or T0-4N2-3)
* Biopsy specimens are available for ER, PgR and Her2 detection, patients should be with triple negative or Her2 positive breast cancer, Her2 positivity is defined as FISH/CISH Her2 positive or IHC Her2 3+, Triple-negative disease defined as negativity for ER, PgR and Her2
* Adequate bone marrow function: Neutrophil ≥ 1.5*109/L; Hb ≥ 100g/L; PLT ≥ 100*109/L
* An estimated life expectancy of at least 12 months
* Willing to take biopsy before neoadjuvant chemotherapy and patients must be accessible for treatment and follow-up
* Women with potential child-bearing must have a negative pregnancy test (urine or serum) within 7 days of drug administration and agree to use an acceptable method of birth control to avoid pregnancy for the duration of the study
* Written informed consent according to the GCP

Exclusion Criteria:

* Prior systemic or loco-regional treatment of breast cancer, including chemotherapy
* Metastatic breast cancer
* With a history of malignant tumor except uterine cervix cancer in situ or skin basal cell carcinoma
* Patients with medical conditions that indicate intolerant to neoadjuvant therapy and related treatment, including uncontrolled pulmonary disease, diabetes mellitis, severe infection, active peptic ulcer, coagulation disorder, connective tissue disease or myelo-suppressive disease
* inadequate liver function (bilirubin > 1.0 times upper normal limit [UNL] and ALT and/or AST> 1.5 UNL associated with alkaline phosphatase > 2.5 UNL; inadequate renal function (creatinine > 1.0 times UNL and in case of limit value, Creatinine clearance < 60 ml/min)
* Contraindication for using dexamethasone
* History of congestive heart failure, uncontrolled or symptomatic angina pectoris, arrhythmia or myocardial infarction; poorly controlled hypertension (systolic BP > 180 mmHg or diastolic BP > 100 mmHg)
* Has peripheral neuropathy ≥ grade 1
* Patient is pregnant or breast feeding
* Known severe hypersensitivity to any drugs in this study
* Treatment with any investigational drugs within 30 days before the beginning of study treatment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-07; Primary Completion 2012-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
pathological complete remission (pCR) rate | after 6 cycles of neoadjuvant therapy

SECONDARY OUTCOMES:
disease free survival (DFS) and overall survival (OS) | 5-year
clinical response rate | after 6 cycles of neoadjuvant therapy
safety profile | during neoadjuvant therapy
breast conservation therapy (BCT) rate | after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kunwei Shen, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (27):
- China (27):
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Guangdong Provincial Maternal and Child Health Hospital, Guangzhou, Guangdong
  - Guangzhou General Hospital of Guangzhou Military Area, Guangzhou, Guangdong
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangyin People's Hospital, Jiangyin, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The Second Affilliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Wujiang First People's Hospital, Wujiang, Jiangsu
  - The third hospital of Nanchang, Nanchang, Jiangxi
  - Linyi People's Hospital, Linyi, Shandong
  - Shanghai Obstetrics and Gynecology Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - the International Peace Maternity and Child health Hospital, Shanghai, Shanghai Municipality
  - Xin Hua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Provincical Cancer Hospital, Taiyuan, Shanxi
  - Fisrt Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Sinkiang Uygur Autonomous Region Cancer Hospital, Ürümqi, Xinjiang
  - Yunnan Provincical Tumor Hospital, Kunming, Yunnan
  - Obstetrics and Gynecology Hospital affiliated to Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Traditional Chinese Medical Hospital, Hangzhou, Zhejiang
  - Ningbo First People's Hospital, Ningbo, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affilliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - Ruian People's Hospital, Wenzhou, Zhejiang

REFERENCES:
- [Background] Yang L, Li LD, Chen YD, Parkin DM. [Time trends, estimates and projects for breast cancer incidence and mortality in China]. Zhonghua Zhong Liu Za Zhi. 2006 Jun;28(6):438-40. Chinese. PMID 17152490
- [Background] Jones SE, Savin MA, Holmes FA, O'Shaughnessy JA, Blum JL, Vukelja S, McIntyre KJ, Pippen JE, Bordelon JH, Kirby R, Sandbach J, Hyman WJ, Khandelwal P, Negron AG, Richards DA, Anthony SP, Mennel RG, Boehm KA, Meyer WG, Asmar L. Phase III trial comparing doxorubicin plus cyclophosphamide with docetaxel plus cyclophosphamide as adjuvant therapy for operable breast cancer. J Clin Oncol. 2006 Dec 1;24(34):5381-7. doi: 10.1200/JCO.2006.06.5391. PMID 17135639
- [Background] Martin M, Pienkowski T, Mackey J, Pawlicki M, Guastalla JP, Weaver C, Tomiak E, Al-Tweigeri T, Chap L, Juhos E, Guevin R, Howell A, Fornander T, Hainsworth J, Coleman R, Vinholes J, Modiano M, Pinter T, Tang SC, Colwell B, Prady C, Provencher L, Walde D, Rodriguez-Lescure A, Hugh J, Loret C, Rupin M, Blitz S, Jacobs P, Murawsky M, Riva A, Vogel C; Breast Cancer International Research Group 001 Investigators. Adjuvant docetaxel for node-positive breast cancer. N Engl J Med. 2005 Jun 2;352(22):2302-13. doi: 10.1056/NEJMoa043681. PMID 15930421
- [Background] Rouzier R, Perou CM, Symmans WF, Ibrahim N, Cristofanilli M, Anderson K, Hess KR, Stec J, Ayers M, Wagner P, Morandi P, Fan C, Rabiul I, Ross JS, Hortobagyi GN, Pusztai L. Breast cancer molecular subtypes respond differently to preoperative chemotherapy. Clin Cancer Res. 2005 Aug 15;11(16):5678-85. doi: 10.1158/1078-0432.CCR-04-2421. PMID 16115903
- See also: published result link — http://www.ncbi.nlm.nih.gov/pubmed/24292815